CLINICAL TRIAL: NCT05822141
Title: Omega-3 Fatty Acid Modulation of Brown Adipose Tissue for Arctic Resilience
Brief Title: Omega-3 Fatty Acids as Regulators of Brown Adipose Tissue During Cold Exposure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tim Mickleborough, Professor of Kinesiology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17715
Record Dates: First submitted 2023-03-27; First posted 2023-04-20 (Actual); Last update posted 2025-04-07 (Actual); Status verified 2025-04

CONDITIONS: Cold Exposure
Keywords: Brown fat; Fish oil; Cold
MeSH Terms: conditions — Common Cold | interventions — Fish Oils

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo controlled, parallel group trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fish Oil (Omega-3 Fatty Acids) (Experimental): 15 subjects will ingest 6 capsules of fish oil of per day for 12 weeks
  Interventions: Dietary Supplement: Fish Oil
- Olive Oil (Placebo Comparator): 15 subjects will ingest 6 capsules of olive oil per day for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fish Oil — For 12 weeks subjects will ingest 6 capsules per day of fish oil (7.8 g/day total omega--3 fatty acids: 3.75 g/day EPA and 1.5 g/day DHA)
  Arms: Fish Oil (Omega-3 Fatty Acids)
Dietary Supplement: Placebo — For 12 weeks subjects will ingest 6 capsules per day of olive oil (each capsule contains 990 mg of olive oil)
  Arms: Olive Oil

SUMMARY:
This clinical trial will assess the whether fish oil supplementation can modulate brown fat activation, shivering, thermal comfort and skin blood flow during cold exposure.

DETAILED DESCRIPTION:
This proof-of-concept study will be conducted as a randomized, double-blind, placebo controlled, parallel group clinical trial in which 30 healthy men and women (ages 18-40 years) will be randomly assigned to fish oil (n=20; 7.8 g/day total n-3 PUFA: 3.75 g/day EPA and 1.5 g/day DHA) or placebo (n=20, olive oil) conditions for 12 weeks. Before beginning supplementation, and at 6- and 12-weeks post-supplementation, whole-body thermoregulation will be assessed by progressively reducing air temperature (from 29°C→4°C, with a wind speed of 4.5 m/s) over a 125-minute period in an environmental chamber. This approach will allow for quantitative determination of fish oil supplementation on body temperature regulation during cold exposure. This approach is novel because it also permits comprehensive assessment of the regulation of core body temperature (rectal temperature) and objective quantification of both autonomic [metabolic heat production (indirect calorimetry), BAT activation (infrared thermography), shivering (accelerometry, electromyography), skin blood flow (laser Doppler)] and behavioral (voluntary control of local thermal comfort) thermoregulatory responses. The advantage of this methodology is that this approach will enable assessment of whether fish oil supplementation is beneficial during exposure to cold environments.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, between the ages of 18 to 40 years.
* Body Mass Index (BMI) of 18.5 to 24.9 kg/m2
* Considered "moderately to highly active" by the International Physical Activity Questionnaire (IPAQ) and the Physical Activity Readiness Questionnaire (PAR-Q+)

Exclusion Criteria:

* History of smoking or recreational smoking, hyperlipidemia, hypertension/cardiovascular disease, diabetes, renal disease, neurological disease, metabolic disease, and bleeding disorders or delayed clotting time.
* Taking SSRI's (antidepressants and anxiety medication), ADD/ADHD medication, and chronically consume pain medication (Aleve, Tylenol, CBD, etc).
* Have or have had chronic disorders of the rectum (e.g., cancer, surgery, active hemorrhoids, etc.) or who currently have related acute conditions (diarrhea, constipation, etc.).
* Have or have had a diagnosis of disorders related to immune suppression and/or autoimmune disease.
* Are pregnant or planning on being pregnant.
* Resting blood pressure of > 130mmHg systolic or 90 mmHg diastolic.
* Resting Pulse rate of > 100 bpm.
* History of regularly consuming fish oil supplements and/or regularly eating more than one fish meal per week.
* Consuming more than one fish meal per week during the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Core Temperature: | 125 minutes
  Core body temperature will be continuously measured by a rectal probe
Metabolic Measurements (indirect calorimetry): | 125 minutes
  Metabolic rate will be measured via indirect calorimetry (i.e., via the analysis of expired gases and ventilation).
Indices of Shivering | 125 minutes
  Surface mechanomyography will be assessed by three triaxial accelerometers adhered to the skin using adhesive tape on the chest, upper back, and thigh will be used to assess shivering
Minnesota Manual Dexterity Test (MMDT) | 10 minutes
  The MMDT [28,29,30] consists of a 60-hole, thin board with red and black blocks (3.7cm) and is comprised of the turning test and the placing test. During the turning test will be modified to only use the dominant hand. During this task, the participant takes a block from the top right corner with their dominant and places it in the hole with their dominant hand. During the placing test, the participant takes one at a time in their dominant hand and places the black in the whole on the board. Scoring of this test is the time it takes to complete each test.
Thermal Perception Scales | 125 minutes
  Thermal perceptions will be assessed using Likert scales for thermal discomfort and thermal sensation. Thermal perceptions will be assessed using Likert scales for thermal discomfort and thermal sensation. Participants will complete Likert scales to assess their thermal comfort (1 = comfortable, 4 = very uncomfortable) and thermal sensation (1 = cold, 4 = neutral, 7 = hot).
Thermal Comfort (behavior) | 125 minutes
  A series of small tubes will be placed on the back of the participant's neck. The participants will control the temperature of the water perfusing these tubes by turning a valve. This will allow for the voluntary control of neck temperatures from 20-35 degrees Celsius. Participants will be instructed to control the temperature of the water bath so that their neck will always be thermally comfortable
Infrared Thermography | 125 minutes
  An infrared thermography camera will be used to measure skin temperature in the supraclavicular (i.e., collar bone) region. This provides a non-invasive estimate of brown adipose tissue activation
Cold Chamber Challenge | 125 minutes
  The environmental chamber set to 29 degrees Celsius (C; 84 degrees Fahrenheit, F) at the beginning of the experimental visit. While in the chamber, participants will be instructed to be sedentary. The chamber will then be cooled at a rate of 1 deg C per 5 minutes until 4 deg C (39.2 deg F) is reached (~125 minutes) with a wind speed of 4.5 m/s. Once 4 deg C air temperature is reached, participants will remain in the chamber for an additional 30 minutes or until the participant can no longer tolerate the cold or if rectal temperature falls below 35.5 deg C (95.9 deg F).
24 Hour Dietary Recalls | 12 weeks
  Participants will be asked to record all food, beverages and supplements consumed during a 24-hour period pre-supplementation, and every 2 weeks during the supplementation period for a total of ~7 dietary recalls to ensure that dietary habits do not change during the 12 week supplementation period.
Skin Temperature | 125 minutes
  Wireless temperature sensors (iButtons, Maxim Inc.) will be attached to 12 sites on the body (forehead, calf, thigh, foot, quadriceps, hamstring, chest, abdomen, upper back, lower back, forearm, and hand) using adhesive tape to measure skin temperature.
Nine Hole Peg Test (NHPT) | 10 minutes
  The NHPT, a manual dexterity test, consists of 9 holes (10mm diameter, 15mm depth) separated by 32mm, and 9 pegs (7mm diameter, 32mm length). During the test, participants will be instructed to take the pegs from a container one by one and place them into the holes on the board as quickly as possible, with their dominant hand. Scoring of this test is the time it takes to complete each test.

SECONDARY OUTCOMES:
Blood Pressure | 10 minutes
  Digital blood pressure cuff will evaluate resting blood pressure
Urine Specific Gravity and Pregnancy Test | 10 minutes
  Hydration status via urine specific gravity (USG) by a handheld refractometer will be utilized and USG < 1.020 will indicate euhydration. For females of child-bearing potential, a small sample of urine will be used for a urine pregnancy test.
Heart Rate | 125 minutes
  Participants will be connected to a 3-lead electrocardiogram (ECG).
Pulse Rate | 10 minutes
  Digital blood pressure cuff will evaluate resting pulse rate
Bone Mineral Density | 10 minutes
  A total-body Dual Energy X-Ray Absorptiometry (DEXA) procedure will be used to assess bone mineral density (g. cm-3) at various body segments (e.g., total body, trunk, hip, leg).
Lean Muscle Mass | 10 minutes
  A total-body Dual Energy X-Ray Absorptiometry (DEXA) procedure will be used to assess lean muscle mass (kilograms or pounds) at various body segments (e.g., total body, trunk, hip, leg).
Fat Mass | 10 minutes
  A total-body Dual Energy X-Ray Absorptiometry (DEXA) procedure will be used to assess fat mass (kilograms or pounds) at various body segments (e.g., total body, trunk, hip, leg).
Body Fat Percentage | 10 minutes
  A total-body Dual Energy X-Ray Absorptiometry (DEXA) procedure will be used to assess body fat percentage (%) at various body segments (e.g., total body, trunk, hip, leg).

CONTACTS AND LOCATIONS:
Overall Officials: Timothy D Mickleborough, PhD, Principal Investigator — Indiana University
Locations (1):
- Human Perfromance Lab, Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No